CLINICAL TRIAL: NCT07135518
Title: Improving Social Climate in Secure Settings With a Compassion Focused Staff Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Psychiatric Clinics Basel (Network)
Responsible Party: Principal Investigator, Andrea Canel, MSc, University Psychiatric Clinics Basel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID ClimACT CFSS
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Social Climate; Compassion; Critical Incident; Staff Support; Workplace Wellbeing
Keywords: Compassion Focused Therapy; Staff Support; Forensic Psychiatry; Social Climate; Workplace Wellbeing; Secure Settings; Staff Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Full CFSS Group (Workshop + Monthly Groups)
  Interventions: Behavioral: Compassion Focused Staff Support
- Partial (Other): Workshop-Only Group
  Interventions: Behavioral: CFT Workshop
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Compassion Focused Staff Support — The Compassion Focused Staff Support (CFSS) intervention is designed to promote emotional resilience, compassion, and affect regulation. The intervention begins with a half-day introductory workshop covering the evolution-informed model of emotion regulation, the three-affect system framework, social mentalities, and the nature of compassion. This workshop provides psychoeducation and experiential exercises to introduce key concepts. Following the workshop, staff participate in six monthly 60-minute team sessions over a six-month period. These sessions involve reflective dialogue, experiential exercises, compassion-focused practices, and group-based exploration of emotionally challenging work situations.
  Arms: Intervention
Behavioral: CFT Workshop — Participants attend a single half-day workshop providing psychoeducation and experiential exercises on compassion, affect regulation, and social mentalities based on Compassion Focused Therapy.
  Arms: Partial

SUMMARY:
This study evaluates the effectiveness of a Compassion Focused Staff Support (CFSS) intervention in improving the social climate of correctional and forensic psychiatric institutions. The intervention is based on Compassion Focused Therapy and designed to support staff in managing stress, enhancing affect regulation, and strengthening compassion toward self and others. Three institutional units are included in the study. One unit is randomly selected to receive the full CFSS intervention, including a half-day introductory workshop and monthly staff support sessions over six months. A second unit serves as a control group and receives no intervention. A third unit receives only the initial workshop without follow-up sessions. The effect of the intervention is evaluated using a pre-test/post-test design. Outcomes include changes in staff-reported and client-reported social climate, assessed with validated questionnaires, as well as institutional data on critical incidents. The study aims to improve working conditions in secure settings and foster more compassionate, effective staff-client interactions.

ELIGIBILITY:
Inclusion Criteria:

Staff Participants:

* Employed at one of the participating correctional or forensic psychiatric units
* Aged 18 years or older
* Willing to provide informed consent

Client Participants:

* Residing in one of the participating correctional or forensic psychiatric units at the time of data collection.
* Aged 18 years or older.
* Capable of providing informed consent

Exclusion Criteria:

Staff Participants:

- None (all eligible staff are invited to participate)

Client Participants:

* Not capable of providing informed consent (e.g., due to acute psychiatric crisis or cognitive impairment).
* Not deemed competent to participate by treatment team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Staff-Perceived Social Climate | T0 (6 months before start of the intervention), T1 (2 weeks before start of the intervention), T2 (2 weeks after last session of the intervention)
  Staff perceptions of social climate will be assessed using the Essen Climate Evaluation Schema (EssenCES), a self-report questionnaire.
Compassion | T0 (6 months before start of the intervention), T1 (2 weeks before start of the intervention), T2 (2 weeks after last session of the intervention)
  Compassionate attitudes and behaviours will be measured using the German version of the Compassionate Engagement and Action Scales (CEAS) to assess staff capacity for self- and other-directed compassion. The CEAS is a self-report questionnaire.

SECONDARY OUTCOMES:
Client-Perceived Social Climate | T0 (6 months before start of the intervention), T1 (2 weeks before start of the intervention), T2 (2 weeks after last session of the intervention)
  Client perceptions of institutional social climate will be measured using the EssenCES. Assessed at three timepoints to evaluate potential parallel changes from the client perspective.
Critical Incidents | T0 (6 months before start of the intervention), T1 (2 weeks before start of the intervention), T2 (2 weeks after last session of the intervention)
  Frequency of critical incidents (e.g., aggression, safety breaches) will be extracted from institutional records. Routinely collected data will be used to assess environmental shifts during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- University Psychiatric Clinics Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No